CLINICAL TRIAL: NCT03361683
Title: Post-extubation High-flow Nasal Oxygen vs. Conventional Oxygen in Patients Recovered From Acute Hypoxemic Respiratory Failure for Preventing Extubation Failure
Brief Title: Post-extubation High-flow Nasal Oxygen for Preventing Extubation Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: REF-1350
Record Dates: First submitted 2017-11-08; First posted 2017-12-05 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-07

CONDITIONS: Extubation Failure
Keywords: High-Flow nasal oxygen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-flow nasal oxygen (Experimental): Randomized patients will receive oxygen through a high flow nasal device capable of delivering humidified, heated air at an output rate of 40 L/min
  Interventions: Device: High-flow nasal oxygen
- Conventional oxygen (Active Comparator): Randomized patients will receive oxygen through a Venturi mask at an air flow of 15 L/min
  Interventions: Device: Venturi mask

INTERVENTIONS:
Device: High-flow nasal oxygen — Randomized patients will receive oxygen through a high nasal flow device capable of delivering humidified, heated air at an output rate of 40 L/min
  Arms: High-flow nasal oxygen
Device: Venturi mask — Randomized patients will receive oxygen through a Venturi mask at an air flow of 15 L/min
  Arms: Conventional oxygen

SUMMARY:
Patients intubated due to acute respiratory failure have a high risk of infectious complications, airway injuries and multiple organic failure, so performing a successful extubation from mechanical ventilation is key. Between 10 and 20% of patients develop extubation failure, which is related to an increased in-hospital death rate, infections, higher costs and longer hospital stays. High-flow nasal oxygen therapy delivers heated, humidified air at flows up to 60L/min, and an oxygen concentration close to 100%, providing a fresh air reservoir at the naseo-pharyngeal level, evening out the peak inspiratory flow rate of the patient, improving air conductance, promoting secretion management, increasing end-expiratory lung volume, and applying a positive end-expiratory pressure. Such effects result in decreased breathing work, dyspnea relief, improved use tolerance, increased oxygenation, and lower fraction of inspired oxygen in patients with hypoxemic respiratory failure. High-flow oxygen therapy has recently been described to decrease extubation failure in a group of patients classified with low failure risk, in comparison to Venturi mask, and it was not inferior to non-invasive mechanical ventilation in high risk patients. However, it is worth pointing out that a large percentage of the patients included in such studies did not develop acute respiratory failure primarily.

Given the beneficial effects described above, the investigators hypothesize that high-flow nasal oxygen therapy decreases the risk of extubation failure in a group of patients that required invasive mechanical ventilation due to primary acute hypoxemic respiratory failure.

DETAILED DESCRIPTION:
Intubated patients recovering from primary acute hypoxemic respiratory failure who have passed a spontaneous breathing trial will be included in the study. Following extubation, patients will be randomized assigned to one of two study groups. Heart rate, breathing rate, median arterial pressure, FiO2, SpO2, and dyspnea and comfort levels will be measured at defined intervals after extubation (basal, 1 hour, 2 hours, 3 hours, 6 hours, 12 hours, 24 hours, and 48 hours). An arterial blood gas test will be performed 60 minutes and 24 hours after extubation. The number of patients fulfilling certain preset criteria regarding extubation failure will be determined.

Extubation failure shall be defined as the need for using invasive mechanical ventilation again within two days following extubation based on the criteria below:

* Breathing rate over 25 breaths per minute for more than two hours.
* Heart rate above 140 beats per minute or with a sustained increase or decrease greater than 20%.
* Clinical data showing fatigue of the respiratory muscles or an increase in breathing work.
* SaO2 <90%; PaO2 <80 mmHg with a FiO2 > 50%.
* Hypercapnia (PaCO2 >45 mmHg or >20% compared to the value before extubation) with a pH below 7.33.

Patients who do not fulfill the extubation failure criteria after the first 48 hours of admission may receive extra supplementary oxygen through any device (e.g., nasal cannula, face mask, reservoir mask, etc.). Every day, SpO2 will be measured and the moment when the patient reaches SpO2 >94% with no need for oxygen will be determined.

ELIGIBILITY:
Inclusion Criteria:

Hypoxemic primary acute respiratory failure

Invasive mechanical ventilation for at least 48 hours

Successful Spontaneous Breathing Trial

Exclusion Criteria:

Immediate indication for invasive mechanical ventilation

Immediate indication for non-invasive mechanical ventilation

Self-extubation

One or more failed Spontaneous Breathing Trial

Chronic respiratory failure

Neuromuscular diseases

Tracheostomy.

Nasal cavity pathology

Facial surgery

Failure to authorize the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Post-extubation failure | First 48 hours
  Number of patients with extubation failure criteria in each group

SECONDARY OUTCOMES:
PaO2/FiO2 Ratio Record. | Post-extubation period and up to 48 hours later.
  An arterial blood gas test will be performed once the high-flow oxygen or Venturi mask is placed.
Determination of FiO2 Requirements. | Post-extubation period and up to 48 hours later.
  Assessment of FiO2 requirements at the time of extubation (when high-flow oxygen or Venturi mask is placed) and then at 60 minutes, 2 hours, 3 hours, 6 hours, 12 hours, 24 hours, and 48 hours. The aim is to maintain SpO2 levels > 94% with the minimal FiO2 possible.
Respiratory Rate Record at Defined Intervals. | Post-extubation period and up to 48 hours later.
  Quantification of respiratory rate at the time of placement high-flow oxygen or Venturi mask and then at 60 minutes, 2 hours, 3 hours, 6 hours, 12 hours, 24 hours and 48 hours.
Heart Rate Record at Defined Intervals. | Post-extubation period and up to 48 hours later.
  Quantification of heart rate at the time of placement high-flow oxygen or Venturi mask and then at 60 minutes, 2 hours, 3 hours, 6 hours, 12 hours, 24 hours and 48 hours.
Mean Arterial Pressure Record at Defined Intervals. | Post-extubation period and up to 48 hours later.
  Quantification of mean arterial pressure at the time of placement high-flow oxygen or Venturi mask and then at 60 minutes, 2 hours, 3 hours, 6 hours, 12 hours, 24 hours and 48 hours.
Treatment Comfort Assessment by means of a Visual Analogue Scale at Defined Intervals. | Post-extubation period and up to 48 hours later.
  To record patient comfort by means of a Visual Analogue Scale tool at the time of placement high-flow oxygen or Venturi mask and then at 60 minutes, 2 hours, 3 hours, 6 hours, 12 hours, 24 hours and 48 hours.
  Visual Analogue Scale range (0 = better to 10 = worse).
Dyspnea Assessment by means of a Visual Analog Scale at Defined Intervals. | Post-extubation period and up to 48 hours later.
  To measure the level of dyspnea by means of a Visual Analogue Scale tool at the time of placement high-flow oxygen or Venturi mask and then at 60 minutes, 2 hours, 3 hours, 6 hours, 12 hours, 24 hours and 48 hours.
  Visual Analogue Scale range (0 = better to 10 = worse).
Number of Days Requiring Oxygen after Successful Extubation | Post-extubation period and up to 14 days later.
  After successful extubation, the level of SpO2 will be measured on a daily basis, recording the time when a level of SpO2> 94% is reached by the patient without the use of supplemental oxygen.
Number of Days Spent in the ICU after Extubation. | Post-extubation period and up to 28 days later.
  There will be quantified the total length of stay in the ICU after extubation.
Days Spent in the Hospital After Extubation. | Post-extubation period and up to 28 days later
  There will be quantified the total length of stay in the hospital after extubation.
Number of Deaths in the ICU after Extubation. | Post-extubation period and up to 28 days later
  There will be quantified the number of patients deceased in each group
Number of Deaths in the Hospital after Extubation. | Post extubation period and up to 28 days later.
  There will be quantified the number of patients deceased in each group

CONTACTS AND LOCATIONS:
Overall Officials: Jose de Jesus Rodriguez-Andoney, MD, Principal Investigator — National Institute of Medical Science and Nutrition Salvador Zubirán
Locations (1):
- National Institute of Medical Science and Nutrition Salvador Zubirán,, México, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chanques G, Constantin JM, Sauter M, Jung B, Sebbane M, Verzilli D, Lefrant JY, Jaber S. Discomfort associated with underhumidified high-flow oxygen therapy in critically ill patients. Intensive Care Med. 2009 Jun;35(6):996-1003. doi: 10.1007/s00134-009-1456-x. Epub 2009 Mar 18. PMID 19294365
- [Result] Dysart K, Miller TL, Wolfson MR, Shaffer TH. Research in high flow therapy: mechanisms of action. Respir Med. 2009 Oct;103(10):1400-5. doi: 10.1016/j.rmed.2009.04.007. Epub 2009 May 21. PMID 19467849
- [Result] Dewan NA, Bell CW. Effect of low flow and high flow oxygen delivery on exercise tolerance and sensation of dyspnea. A study comparing the transtracheal catheter and nasal prongs. Chest. 1994 Apr;105(4):1061-5. doi: 10.1378/chest.105.4.1061. PMID 8162725
- [Result] Ricard JD. High flow nasal oxygen in acute respiratory failure. Minerva Anestesiol. 2012 Jul;78(7):836-41. Epub 2012 Apr 24. PMID 22531566
- [Result] Groves N, Tobin A. High flow nasal oxygen generates positive airway pressure in adult volunteers. Aust Crit Care. 2007 Nov;20(4):126-31. doi: 10.1016/j.aucc.2007.08.001. Epub 2007 Oct 10. PMID 17931878
- [Result] Corley A, Caruana LR, Barnett AG, Tronstad O, Fraser JF. Oxygen delivery through high-flow nasal cannulae increase end-expiratory lung volume and reduce respiratory rate in post-cardiac surgical patients. Br J Anaesth. 2011 Dec;107(6):998-1004. doi: 10.1093/bja/aer265. Epub 2011 Sep 9. PMID 21908497
- [Result] Spence KL, Murphy D, Kilian C, McGonigle R, Kilani RA. High-flow nasal cannula as a device to provide continuous positive airway pressure in infants. J Perinatol. 2007 Dec;27(12):772-5. doi: 10.1038/sj.jp.7211828. Epub 2007 Aug 30. PMID 17762844
- [Result] Chidekel A, Zhu Y, Wang J, Mosko JJ, Rodriguez E, Shaffer TH. The effects of gas humidification with high-flow nasal cannula on cultured human airway epithelial cells. Pulm Med. 2012;2012:380686. doi: 10.1155/2012/380686. Epub 2012 Sep 3. PMID 22988501
- [Result] Sreenan C, Lemke RP, Hudson-Mason A, Osiovich H. High-flow nasal cannulae in the management of apnea of prematurity: a comparison with conventional nasal continuous positive airway pressure. Pediatrics. 2001 May;107(5):1081-3. doi: 10.1542/peds.107.5.1081. PMID 11331690
- [Result] Roca O, Riera J, Torres F, Masclans JR. High-flow oxygen therapy in acute respiratory failure. Respir Care. 2010 Apr;55(4):408-13. PMID 20406507
- [Result] Maggiore SM, Idone FA, Vaschetto R, Festa R, Cataldo A, Antonicelli F, Montini L, De Gaetano A, Navalesi P, Antonelli M. Nasal high-flow versus Venturi mask oxygen therapy after extubation. Effects on oxygenation, comfort, and clinical outcome. Am J Respir Crit Care Med. 2014 Aug 1;190(3):282-8. doi: 10.1164/rccm.201402-0364OC. PMID 25003980
- [Result] Lenglet H, Sztrymf B, Leroy C, Brun P, Dreyfuss D, Ricard JD. Humidified high flow nasal oxygen during respiratory failure in the emergency department: feasibility and efficacy. Respir Care. 2012 Nov;57(11):1873-8. doi: 10.4187/respcare.01575. Epub 2012 Mar 13. PMID 22417844
- [Result] Hernandez G, Vaquero C, Gonzalez P, Subira C, Frutos-Vivar F, Rialp G, Laborda C, Colinas L, Cuena R, Fernandez R. Effect of Postextubation High-Flow Nasal Cannula vs Conventional Oxygen Therapy on Reintubation in Low-Risk Patients: A Randomized Clinical Trial. JAMA. 2016 Apr 5;315(13):1354-61. doi: 10.1001/jama.2016.2711. PMID 26975498
- [Result] Hernandez G, Vaquero C, Colinas L, Cuena R, Gonzalez P, Canabal A, Sanchez S, Rodriguez ML, Villasclaras A, Fernandez R. Effect of Postextubation High-Flow Nasal Cannula vs Noninvasive Ventilation on Reintubation and Postextubation Respiratory Failure in High-Risk Patients: A Randomized Clinical Trial. JAMA. 2016 Oct 18;316(15):1565-1574. doi: 10.1001/jama.2016.14194. PMID 27706464